CLINICAL TRIAL: NCT03201484
Title: Patient Reported Outcomes Following Parotid Resections: Version 2
Brief Title: Patient Reported Outcomes Following Parotid Resections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 221947
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Parotidectomy, Patient-reported Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: FACE-Q questionnaire, 3D photography — FACE-Q questionnaire, 3D photography

SUMMARY:
A study correlating patient reported outcomes measured by a validated tool with physical measurements recorded by 3d photography of patients undergoing parotid resections

DETAILED DESCRIPTION:
The studies primary aim is to use the FACE-Q (a validated patient reported outcome (PRO) scale) for patients undergoing parotidectomy to subjectively measure the functional and aesthetic impact of the surgery1. It is hypothesized that patients undergoing parotidectomy have long-standing under-reported functional and cosmetic issues. Currently most parotid defects are not reconstructed. A secondary aim is to objectively analyse the volume of the parotid gland pre- and post-operatively to guide reconstructive surgery in patient with parotid tumours.

Head and neck tumours are common. Most salivary gland tumours arise from the parotid gland and 80% are benign. Tumour resection can be limited/partial, superficial, total or radical depending upon the pathology2. This can lead to a cosmetic deformity in the pre-auricular /cheek region, infra-auricular region causing a superior cervical depression (especially if combined with a neck dissection) and retromandibular regions2,3. More than 50% of patients report being affected by facial contour abnormalities after parotidectomy and their deformity can be both visible on direct and lateral facial views4. The cosmetic defect following parotidectomy has been rated from moderate to severe disgurement5. Facial disfigurement experienced by head and neck cancer patients has a strong impact on their quality of life6,7 (both in function and cosmesis). This is accentuated by the central role of the face in social communication and expression. Despite these facts there is little evidence on PRO measures post parotidectomies.

PRO's are essential in current medical practice to view success of an intervention from a patient's perspective. Two types of questionnaires are available- generic (e.g. SF-36) and disease specific (e.g. FACE- Q). Generic assess the disease effect on the whole person irrespective of the medical condition. Disease specific assess interventions in a particular disease. They are more sensitive to detect changes due to focused questions. The FACE-Q questionnaire is a recently designed gold standard PRO that is disease specific. The FACE-Q measures 4 domains- satisfaction with facial appearance, adverse effects (both of these highlight the effects on a specific facial area e.g. lips, eye etc), health-relate quality of life and process of care (both of these are relevant to al facial patients). It achieves this as it has over 40 scales each with a series of questions around one central concept. Patient responses are graded on a 4 point scale and then converted to a score on a scale from 0-100. A higher score means improved quality of life. There is no overall score, only scores for each independent scale. As scales are independent only the scales most relevant to a specific research objective or patient population need be administered. Patients can complete the questionnaire pre and post operatively to view the impact of the intervention. An advantage is that it only takes a few minutes to complete. The dis-advantage of the FACE-Q could be perceived that it was initially developed for aesthetic facial procedures however the questions are directly applicable for reconstructive facial procedures. Also research is still undergoing regarding the clinical meaning/clinical significance of the FACE-Q but it still allows PRO quantitative data pre and post procedure to aid evaluation

There is little reconstruction post parotidectomy. However, the goals of reconstruction are both functional (e.g. management of weakness of the lower lip or oral continence, reconstruction of the facial nerve and prevention of Gustatory sweating) and aesthetic2. A few possible methods have been described for reconstruction. Primary reconstruction of small defects are usually with local fascial flaps2 e.g. SMAS flaps5 and large defects with muscle flaps2 e.g. Sternocleidomastoid8. Secondary reconstruction involves fat grafting5 or correction of lip asymmetry. The main method of reconstruction involves the defect being analysed and subjectively "compared" to the contralateral side2. Recent papers have attempted to improve accuracy. Some have reported abnormal volumes i.e. tumour size. However, they have not reported normal volumes (i.e. size of defect)5.MRI has been used to measure volume of defects left behind, however this is not totally accurate as it only measured the largest transverse dimension and requires further expensive imaging5. Therefore to improve outcomes improved accuracy on the dimensions of the defect is required before reconstruction.

Furthermore, although some reconstruction outcomes have been measured by subjective methods8, there is none by a validated questionnaire e.g. the FACE-Q. End points such as morbidity and mortality and recurrence rates are only one measure of treatment success. In addition, there are few objective outcomes reported e.g. using a visual analogue scale9 has been mentioned but this is less accurate than using pre and post op 3D photography.

This study will look at prospective analysis of 50 consecutive patients undergoing parotidectomy by consultant head and neck surgeons (ENT and maxillofacial surgeons) at 1 academic tertiary centre (Guy's Hospital). A range of adults from 18-80 years old with capacity and of any gender or ethnicity will be assessed. Patients having both benign and malignant parotid resection with either partial or superficial or total parotidectomy or neck dissection will be included. Data to be collected includes pre-operative FACE-Q analysis and non-invasive 3D camera measurements, demographic data, tumour pathology, tumour size, defect size, postoperative radiation and duration of follow-up. Follow up will be from 3 months up to 1 year post surgery using the FACE-Q and a non-invasive 3D camera.

There is no obvious risk to the patient as a validated questionnaire will be used and a non-invasive investigation tool. The patient will not be subject to any extra treatment or time in hospital for this particular group of patients.

No previous trials have been performed that are relevant to this study.

ELIGIBILITY:
Inclusion Criteria:

- Adults 18-80 years old. Any gender. Any ethnicity. Capacity to participate in the study. Patients having both benign and malignant parotid tumours for resection including having a neck dissection.

Patients having both primary superficial or total parotidectomy.

Exclusion Criteria:

* Children (< 18 years old). Adults > 80 years old i.e. too old for surgery/follow up Patients without capacity. Primary parotid surgery (not secondary procedures). Patients having radical parotidectomy with additional facial nerve sacrifice. Patients have immediate reconstruction (e.g. with free flap). Previous/current facial surgery/co-morbidity e.g. facial palsy Co-morbidity precluding surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will look at prospective analysis of 50 consecutive patients undergoing parotidectomy by consultant head and neck surgeons (ENT and maxillofacial surgeons) at 1 academic tertiary centre (Guy's Hospital). It is expected all patients will be recruited within 1 year (based on previous hospital data). A range of adults from 18-80 years old and of any gender or ethnicity will be recruited from the Head and Neck cancer MDT clinic. Patients having both benign and malignant parotid resection with either partial or superficial or total parotidectomy or neck dissection will be included. Data to be collected includes pre-operative FACE-Q analysis and non-invasive 3D camera measurements, demographic data, tumour pathology, tumour size, defect size, postoperative radiation and duration of follow-up. Follow up will be from 6 weeks up to 1 year post surgery using the FACE-Q and a non-invasive 3D camera. No previous trials have been performed that are relevant to this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes as measured by the validated FACE-Q questionnaire | 1 year
  Patient Reported Outcomes as measured by the validated FACE-Q questionnaire
Physical cheek defect as measured with 3D photography | 1 year
  Patient Reported Outcomes as measured by the validated FACE-Q questionnaire